CLINICAL TRIAL: NCT01511471
Title: Ticagrelor in Clopidogrel Resistant Patients Undergoing Chronic Hemodialysis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Patras (Other)
Responsible Party: Principal Investigator, Dimitrios Alexopoulos, Clinical Professor, University of Patras
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: PATRASCARDIOLOGY-9
Record Dates: First submitted 2012-01-12; First posted 2012-01-18 (Estimated); Last update posted 2012-02-03 (Estimated); Status verified 2012-02

CONDITIONS: Platelet Reactivity
Keywords: Ticagrelor; platelet reactivity; clopidogrel; haemodialysis
MeSH Terms: interventions — Ticagrelor

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ticagrelor (Experimental): Ticagrelor 90mg twice a day for 15 days
  Interventions: Drug: Ticagrelor

INTERVENTIONS:
Drug: Ticagrelor — Ticagrelor 90mg twice a day for 15 days

SUMMARY:
Clopidogrel administration is commonly prescribed in patients undergoing percutaneous coronary intervention, in patients with previous stroke and in patients under chronic hemodialysis via fistulae. Patients with chronic renal failure present lower clopidogrel response compared to those with normal renal function. Ticagrelor is a new oral direct-acting antagonist, which provides greater platelet inhibition in both clopidogrel responders and non-responders. It has also been shown that in patients with chronic kidney disease (creatinine clearance <60 mL/min)ticagrelor achieved an absolute risk reduction of cardiovascular death, myocardial infarction, and stroke greater than that of patients with normal renal function. Clopidogrel resistant patients as assessed by VerifyNow P2Y12(Accumetrics)will be administered after informed consent ticagrelor 90 mg twice daily for 15 days. Platelet reactivity will be determined at the end of the treatment period. Bleeding events, major adverse cardiac events and any side effects until Day 15 will be reported in a descriptive manner.

ELIGIBILITY:
Inclusion Criteria:

* Age≥18 years
* Chronic renal failure under haemodialysis
* Platelet reactivity under clopidogrel 75mgx1 ≥235 PRU
* Informed written consent

Exclusion Criteria:

* Recent (within 1 month) PCI or ACS
* Requirement for oral anticoagulant prior to the Day 14 visit
* PLTs<100.000 / μL), Hct <28%, Hct > 52% at randomization
* Increased risk of bradycardiac events.
* Severe uncontrolled chronic obstructive pulmonary disease
* Known severe hepatic impairment
* History of gastrointestinal bleeding, genitourinary bleeding or other site abnormal bleeding within the previous 6 months.
* Other bleeding diathesis, or considered by investigator to be at high risk for bleeding
* Concomitant therapy with a strong cytochrome P-450 3A inhibitor or inducer
* Recent (<6weeks)major surgery including CABG
* Recent (<6weeks)stroke or any prior intracranial bleeding

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-01; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Platelet reactivity assessed by VerifyNow P2Y12 assay | Day 15

SECONDARY OUTCOMES:
Bleeding events according to TIMI criteria | Day 15
  Major, minor or minimal bleeding events according to TIMI criteria
Major adverse cardiovascular events | Day 15
  Death, non-fatal myocardial infarction and stroke

CONTACTS AND LOCATIONS:
Locations (2):
- Greece (2):
  - Agios Andreas General Hospital, Nephrology Department, Pátrai, Achaia
  - Cardiology Department Patras University Hospital, Rio, Achaia